CLINICAL TRIAL: NCT04518579
Title: Effect of Epidural-inhalational Versus Epidural-intravenous Anaesthesia on Anti-tumor Immunity in Patients Undergoing Open Surgery for Cancer Colon
Brief Title: Epidural-inhalational Versus Epidural-intravenous Anaesthesia on Anti-tumor Immunity in Patients With Cancer Colon
Acronym: tumorimmunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Bahaa Gamal, Assistant lecturer, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 375
Record Dates: First submitted 2020-08-09; First posted 2020-08-19 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Immunity Factors in Cancer Colon Patients
MeSH Terms: interventions — Tea

STUDY DESIGN:
Intervention Model Description: Group (EP) received epidural - propofol based anesthetic technique and postoperative analgesia through patient controlled epidural analgesia and Group (EH) received epidural- inhalational based anesthetic technique and postoperative analgesia through patient controlled epidural analgesia
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (EP) (Active Comparator): Group (EP) received epidural (fentanyl and bupivacaine) - propofol based anesthetic technique and postoperative analgesia through patient controlled analgesia device (PCA)
  Interventions: Procedure: thoracic epidural
- Group (EH) (Active Comparator): Group (EH) received epidural (fentanyl and bupivacaine)- inhalational based anesthetic technique and postoperative analgesia through patient controlled analgesia device (PCA)
  Interventions: Procedure: thoracic epidural

INTERVENTIONS:
Procedure: thoracic epidural — undergo insertion of an epidural catheter, between T9 and T11 in patients undergoing left-sided resections and between T8 and T10 in patients undergoing right-sided resections
  Other Names: thoracic epidural catheter

SUMMARY:
Surgery is the primary treatment for colon cancer. However, the rate of recurrence or metastasis in colon cancer can be as high as 30%, even in stages 1 and 2 . Most colon cancer-related deaths are caused by metastatic disease . Many patients with colon cancer harbour micrometastases and disseminated tumour cells at the time of surgery . Whether the micrometastases develop into clinically significant metastases depends on the immune system's ability to eradicate them.The aim of the study is to declare the effect of epidural-intravenous based anesthetic technique on anti-tumor immunity and in comparison to epidural inhalational based anesthetic technique in patients undergoing open surgical resection of colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 yrs.
* ASA class I and II
* Elective open surgery for non-metastatic cancer colon stage I,II

Exclusion Criteria:

* Patient refusal
* Known allergy to the study medications
* Patients with compromised immune function ( associated blood diseases, immunosuppressive drugs, chemotherapeutic agents, corticosteroids)
* Contraindications to epidural insertion e.g. infection at insertion site and coagulopathy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
anti tumour immunity | preoperative and Day 1 postoperatively
  Venous blood samples are withdrawn. Samples for measurement of percentage of expression of CD8,CD16 and CD56 will be collected in sodium heparin anticoagulant tubes and will be processed according to manufacturer's instructions,and samples for VEGF-C will be centrifuged at 4000 g. Thereafter, the serum will be stored at -22 C for future measurement

SECONDARY OUTCOMES:
change in pain intensity | 24 hours postoperative
  pain intensity measured by Visual analogue scale from 0 to 10 where 0 no pain and 10 is sever pain

CONTACTS AND LOCATIONS:
Overall Officials: samy ab amr, professor, Study Chair — dean of SECI
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No